CLINICAL TRIAL: NCT02527941
Title: Effect of Bacterial Vaginosis and Its Treatment on HIV Susceptibility and Female Genital Immunology
Brief Title: Effect of Bacterial Vaginosis on HIV Susceptibility and Female Genital Immunology
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Rupert Kaul, Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UTorontoBV
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Bacterial Vaginosis; HIV Infections
Keywords: Genital immunology; HIV susceptibility; Microbiome; Bacterial vaginosis; Virus entry assay
MeSH Terms: conditions — Vaginosis, Bacterial; HIV Infections | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- metronidazole (Experimental): 50 women who test negative for HIV and classical sexually transmitted infections but test positive for Bacterial Vaginosis will be treated with metronidazole at a dosage of 400mg/dose, 3 doses per day, for 7 days (as per Kenyan National Guidelines).
  Interventions: Drug: Metronidazole

INTERVENTIONS:
Drug: Metronidazole — Participants will be provided with oral metronidazole 400mg po tid for one week, and followed up one month after treatment initiation.
  Other Names: flagyl

SUMMARY:
A non-randomized, interventional, longitudinal clinical study to quantify the impact of bacterial vaginosis treatment on HIV susceptibility and genital immunology in Kenyan women.

DETAILED DESCRIPTION:
Bacterial Vaginosis (BV), defined as an alteration in the normal vaginal bacteria ("microbiome"), is characterized by a reduction of hydrogen peroxide-producing gram-positive lactobacilli and overgrowth of gram-negative and anaerobic bacteria. BV is more prevalent in SSA and usually recurs soon after treatment. BV is associated with vaginal inflammation, an increased HIV acquisition risk among uninfected women, and increased HIV transmission to the male sexual partner of a co-infected woman. Therefore, BV may be responsible for up to 17% of HIV transmission events in SSA.

There are several hypotheses for the mechanisms by which BV may increase the risk of HIV acquisition. These include the disruption of mucosal barrier, alteration of protective innate immunity, and increased number and/or susceptibility of HIV target cells in the genital mucosa. Longitudinal studies that address the mechanisms by which the vaginal microbiota alters host mucosal immunology and HIV risk will help us better understand the impact of BV and it's treatment on mucosal immunology and HIV susceptibility. The goal of this non-randomized, interventional, longitudinal clinical study is to use a novel ex vivo HIV infectivity assay developed in the Kaul lab to quantify the effect of BV and its treatment on HIV susceptibility and genital immunology in HIV-uninfected women from Nairobi, Kenya. Fifty HIV, STI-uninfected women with bacterial vaginosis on Nugent scoring will be provided with one week of metronidazole 400mg po three times daily (as per Kenyan National Guidelines). Cytobrush and vaginal SoftCup sampling will be performed at baseline and 4 weeks after treatment initiation, at the same stage of the menstrual cycle. The primary endpoint will be pseudovirus entry into cervix-derived CD4+ T cells. Secondary endpoints will include a pre-defined cervico-vaginal inflammation score; genital CD4+ T cell immune characteristics; the genital microbiome; the genital proteome.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are over 18 years of age, not pregnant and willing to give informed consent, and answer short questionnaires on economic status, and sexual risk behavior.
2. Willing to comply with the requirements of the protocol
3. HIV and classical STI (see below) negative
4. test positive for BV, defined as Nugent score from 7-10
5. willing to take oral metronidazole twice a day for 7 days
6. willing to abstain from alcohol during and for 48 hours after metronidazole treatment

Exclusion Criteria:

1. HIV infected
2. Deemed by physician to be unlikely to complete study protocol.
3. Pregnant.
4. Irregular menstrual cycle, or actively menstruating at the time of genital sampling.
5. Tested positive for classical STIs or having genital ulcers
6. Prior hysterectomy
7. Contraindication, allergy or intolerance to use of metronidazole

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percent HIV pseudovirus entry into cervical CD4+ T cells. | up to 8 months
  The percentage of cervical CD4+ T cells per cytobrush infected ex vivo by an HIV pseudovirus construct will be quantified by flow cytometry.
Total number of cervical CD4+ T cells infected ex vivo with HIV. | up to 8 months
  The total number of cervical CD4+ T cells per cytobrush infected ex vivo by an HIV pseudovirus construct will be quantified by flow cytometry.

SECONDARY OUTCOMES:
A genital inflammation score based on genital levels of pro-inflammatory cytokines and chemokines. | up to 8 months
  Level of 14 genital cytokines/chemokines (GM-CSF, IL-1a, IL-8, MCP-1, MIG, MIP-3a, RANTES, IL-10, IL-17, IL-1b, IL-6, IP-10, MIP-1b, TNF-a) will be combined into a genital inflammation score [Arnold K et al, Muc Immunol, 2015].
The cervico-vaginal microbiome. | up to 8 months
  The cervico-vaginal microbiome will be assessed by 16s rRNA sequencing before and after metronidazole therapy.
Genital proteome analysis. | up to 8 months
  The genital proteome will be assessed by mass spectroscopy before and after metronidazole therapy.
CD4+ expression of pre-defined HIV susceptibility markers | up to 8 months
  Surface expression of CCR5, CD69, a4b7 and a4b1 by endocervical CD4 T cells before and after metronidazole therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Kaul, MD/PhD, Principal Investigator — University of Toronto
Locations (1):
- Kenya AIDS Vaccine Initiative Clinic, Nairobi, Kenya